CLINICAL TRIAL: NCT06498999
Title: Development and Validation of a 4-STEP-Training Program for Social Media Addiction (4-STEP-TPS) Among Young Adults: A Randomized Control Trial
Brief Title: 4-STEP-Training Program for Social Media Addiction (4-STEP-TPS) Among Young Adults
Acronym: 4-STEP-TPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Government College University Faisalabad (Other)
Responsible Party: Principal Investigator, Qasir Abbas, Assistant Professor - Clinical Psychology, Government College University Faisalabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCUF
Record Dates: First submitted 2024-07-01; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Social Media Addiction
Keywords: Training Program; 4-STEP-Training Program for Social Media Addiction; Social Media Addiction; Social Networking; Flourishing; Dysfunctional Patterns; Fatigue Assessment Scale (FAS); Intervention
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Intervention Model Description: A randomized control trial design will be used in this study. It will be a three-arm study with the following groups: (1) an experimental group receiving the intervention in a group setting, (2) an experimental group receiving the intervention in an individual setting, and (3) a waitlist control group. In this research, a parallel group design will be used, with treatment given to all participants in a parallel manner. The allocation ratio and framework will be equivalence, meaning that each of the three groups will have an equal number of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group: Individual Setting (Experimental): 4-STEP-Training Program in 1-1 Setting
  Interventions: Behavioral: 4-STEP-Training Program for Social Media Addiction (4-STEP-TPS)
- Experimental Group: Group Setting (Experimental): 4-STEP-Training Program in Group Setting
  Interventions: Behavioral: 4-STEP-Training Program for Social Media Addiction (4-STEP-TPS)
- Control Group (No Intervention): No Intervention

INTERVENTIONS:
Behavioral: 4-STEP-Training Program for Social Media Addiction (4-STEP-TPS) — 4 Modules with 1 Module being delivered in 1 weekly session of approximately 90 minutes. The details of each module/step is described as follows:
  Step 1 (Module 1): S = Screening, Assessment and Psychoeducation: Involves screening and assessment of the problem, interpretation of the results, feedback and psychoeducation, identifying and breaking the resistance, motivation, and conceptualization.
  Step 2 (Module 2): T = Treatment Conceptualization and Planning: Involves pattern identification, distortion identification, as well as pattern and distortions modifications.
  Step 3 (Module 3): E = Effective Management Strategies: Involves management strategies to treat the earlier identified patterns as well as the implementation and confirmation of activities via a Pattern Schedule Chart.
  Step 4 (Module 4): P = Prevention (Lapse-Relapse): Involves self-reflection and support building, monitoring and dependency check and slip plans and support additions
  Arms: Experimental Group: Group Setting; Experimental Group: Individual Setting

SUMMARY:
The goal of this clinical trial is to develop a comprehensive Training Program intervention for social media addiction called the 4-STEP-Training Program for Social Media Addiction (4-STEP-TPS) and to learn if the 4-STEP-TPS will address and help manage the problems related to social media addiction. Other key objectives include the management of dysfunctional patterns, the promotion of positive patterns and healthy lifestyle, and the promotion of daily life activities and productivity.

Young Adult participants will take the 4-week 4-STEP-TPS Program with 1 weekly session in either individual or group settings or be placed on a waitlist control.

DETAILED DESCRIPTION:
Participants In this research, a sample of N=400 young adults will be initially enrolled for eligibility screening assessment from all over Pakistan using purposive sampling techniques. The participants' age range will be 18-30 years having no physical/psychiatric/psychological conditions. N=90 participants after the eligibility assessment and screening will be allocated to experimental and waitlist treatment condition.

Expected Outcomes This study will provide valuable information to the mental health practitioners to treat and develop the guidelines and protocol for young adults with social media addiction. This 4-STEP-Training Program will provide understanding and insight to the participants about the problems related to social media addiction. Further, this training program will address the dysfunctional patterns associated with social media addiction, including FoMO and phubbing, as well as fatigue, insomnia, and psychological distress. Moreover, this training program will improve participants' productivity and flourishing while significantly reducing the level of social media addiction.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18-30 years
* No physical, psychiatric, or psychological conditions
* Minimum score of 84 on the Social Networking Addiction Scale (SNAS)
* Minimum score of 60 on the Secure Flourish Index (SFI)

Exclusion Criteria:

* Age below 18 or above 30 years
* Presence of any physical, psychiatric, or psychological conditions
* Score below 84 on the Social Networking Addiction Scale (SNAS)
* Score below 60 on the Secure Flourish Index (SFI)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Social Networking Addiction Scale (SNAS) | At screening, after 4 weeks, and reassessment up to 6 months
  The Social Networking Addiction Scale (SNAS) was developed to measure addiction of all forms of social networking across six-dimensions salience (items 1-4), mood modification (items 5-7), tolerance (items 8-10), withdrawal (items 11-14), conflict (item 15-17), and relapse (items 18-21) (Shahnawaz & Rehman, 2020). The SNAS is a self-reported scale which entails 21-items scale rated on 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). The score can range from 21 to 147. Any score above a total score of 84 signifies addiction. The scale has demonstrated good test-retest reliability of 0.88 and good validity as reported by Shahnawaz and Rehman (2020).
Secure Flourish Index (SFI) | At screening, after 4 weeks, and reassessment up to 6 months
  The Secure Flourish Index (SFI) was developed to measure long-term flourishing across 6 domains happiness and life satisfaction (items 1-2), physical and mental health (items 3-4), meaning and purpose (items 5-6), character and virtue (items 7-8), close social relationships (items 9-10), and financial and material stability (items 11-12) (Weziak-Bialowolska et al., 2017). It is a self-report scale with 2 items for each of the 6 domains, totaling to 12 items rated on a scale of 0-10. Total scores range from 0 to 120 with higher scores indicating greater flourishing. It has an internal consistency of 0.85 and good construct validity (Weziak-Bialowolska et al., 2017).
Fear of Missing Out Scale (FoMOs) | At screening, after 4 weeks, and reassessment up to 6 months
  The Fear of Missing out Scale (FoMOs) was developed to measure FoMO (Przybylski et al., 2013). It is a self-report questionnaire of 10-items rated on a 5-point Likert scale ranging from 1 (not at all true of me) to 5 (extremely true of me). The total scores of the scale range between 10 and 50, where higher scores indicate a higher level of fear of missing out. The scale has been shown to exhibit strong internal consistency of 0.87 to 0.90 and good validity (Przybylski et al., 2013).
Pubbing Scale (PS) | At screening, after 4 weeks, and reassessment up to 6 months
  The Phubbing Scale was developed to measure the phubbing behaviors (Karadağ et al., 2015). The scale contains 10 items, rated from 1 (never) to 5 (always) in a 5-point Likert scale, the following 2 factors were found: (i) Factor 1 (1-5 items; α = .87) and (ii) Factor 2 (6-10 items; α = .85). The content of these factors can be summarized as follows:
  (i) Communication disturbance: Higher scores indicate that participants often disturb their existing communications by dealing with their mobile phones in a face-to-face communication environment.
  (ii) Phone obsession: Higher scores indicate that participants constantly need their mobile phone in environments lacking face-to-face communication.
Fatigue Assessment Scale (FAS) | At screening, after 4 weeks, and reassessment up to 6 months
  The Fatigue Assessment Scale (FAS) was developed to evaluate the physical and mental symptoms of fatigue (Michielsen et al., 2003). It is a self-report measure with 10 items rated on a 5-point Likert scale ranging from 1 (never) to 5 (always). The scale has 2 subscales, with mental fatigue measured by the sum of items 3, 6, 7, 8, and 9 and physical fatigue measured by the sum of items 1, 2, 4, 5 and 10. Items 4 and 10 are reverse-scored. The total scores range from 10, indicating the lowest level of fatigue, to 50, indicating the highest level of fatigue. The scale has an internal consistency of 0.90 and good validity (Michielsen et al., 2003).
Insomnia Severity Index (ISI) | At screening, after 4 weeks, and reassessment up to 6 months
  The Insomnia Severity Index (ISI) was developed as a screening measure for insomnia as well as an outcome measure in treatment research (Bastien et al., 2001). It is a self-report measure with 7 items rated on a 5-point Likert scale ranging from 0 to 4. The total scores range from 0 to 28, with higher scores indicating more acute insomnia symptoms. Although not validated, the developers suggest cutoff scores to be used for interpretation, with total scores of 0-7 indicating "no clinically significant insomnia," scores between 8-14 indicating "subthreshold insomnia," scores between 15-21 indicating "clinical insomnia (moderate severity)," and scores in the range 22-28 indicating "clinical insomnia (severe)." The scale has an internal consistency of 0.74 (Bastien et al., 2001).
Depression, Anxiety and Stress Scales (DASS) | At screening, after 4 weeks, and reassessment up to 6 months
  The DASS-21 is the shortened version of the DASS-42 was designed to measure the symptoms of depression, anxiety, and stress (Lovibond & Lovibond, 1995). It is a self-report measure with 21 items rated on a 4-point Likert scale ranging from 0 to 3. Each of the three DASS-21 scales depression (items 3, 5, 10, 13, 16, 17, 21), anxiety (items 2, 4, 7, 9, 15, 19, 20), and stress (items 1, 6, 8, 11, 12, 14, 18) contains 7 items. The scale has good internal consistency and construct validity in both clinical and non-clinical samples (Antony et al., 1998). Scores on the DASS-21 will need to be multiplied by 2 to calculate the final score. After obtaining the final score for each depression, anxiety, and stress, the final score is compared to the recommended cut-off scores for severity levels (normal, moderate, severe).

CONTACTS AND LOCATIONS:
Overall Officials: Qasir Abbas, PhD, Principal Investigator — Assistant Professor - Clinical Psychology
Locations (1):
- Government College University Faisalabad, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No